CLINICAL TRIAL: NCT02283099
Title: An Open Label, Single Center, Dose Escalation Phase I Trial to Assess the Safety, Tolerability and Immunogenicity of a Single Ascending Dose of the Ebola Virus Vaccine rVSVΔG-ZEBOV-GP (BPSC1001)
Brief Title: Phase I Trial to Assess the Safety, Tolerability and Immunogenicity of a Ebola Virus Vaccine (rVSVΔG-ZEBOV-GP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Center for Infection Research (Other); Philipps University Marburg (Other); World Health Organization (Other); Clinical Trial Center North (Unknown); University Hospital, Geneva (Other); Albert Schweitzer Hospital (Other); Institute of Tropical Medicine, University of Tuebingen (Other); Wellcome Trust (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKE-DZIF2-VSV{Delta}G/ZEBOVGP
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Ebola virus, vaccination, phase I, healthy volunteers
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rVSVΔ-ZEBOV-GP (BPSC1001) (Experimental): Subjects will be allocated to three cohorts of 10 subjects each receiving one single vaccine injection administered as an i.m. injection.
  Interventions: Biological: rVSVΔ-ZEBOV-GP

INTERVENTIONS:
Biological: rVSVΔ-ZEBOV-GP — single dose of rVSVΔ-ZEBOV-GP (3x10^6 pfu, 2x10^7 pfu or 3x10^5)
  Other Names: BPSC1001

SUMMARY:
The study is designed to establish safety, tolerability and immunogenicity of rVSVΔG-ZEBOV-GP (BPSC1001), an Ebola Virus Vaccine candidate (recombinant vesicular stomatitis virus (VSV) expressing the envelope glycoprotein of Ebola Virus Zaire), investigated at three different dose levels in 30 healthy adults in Germany. This study is part of the WHO led VEBCON consortium that is aiming to generate harmonized data for the rVSVΔG-ZEBOV-GP (BPSC1001) vaccine candidate to allow optimized rapid decisions on dose and safety.

DETAILED DESCRIPTION:
This study is being conducted to assess safety and immunogenicity of an experimental ebola vaccine.

An outbreak due to the Ebola Zaire (ZEBOV) strain of unprecedented magnitude and scope and with a high mortality continues to spread across West Africa. No vaccine is currently licensed.

The specific opportunity at hand with rVSVΔG-ZEBOV-GP (BPSC1001) is to achieve long-lasting protective immunity to ZEBOV on a time scale of weeks in humans upon a single-shot vaccination, offering a discrete benefit over prime-boost vaccination protocols. The current outbreak represents a global health emergency and the need for access to therapeutic intervention and vaccines is paramount.

The vaccine investigated in this study might provide a critical tool to suppress future out-breaks of EVD in areas at risk.

This study is 1 of 4 clinical trials currently conducted as part of the WHO-led VEBCON consortium, aiming to generate harmonized data for the rVSVΔG-ZEBOV-GP (BPSC1001) vaccine candidate to allow optimized rapid decisions on dose and safety.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the subject information and to personally sign the informed consent
* Provided written informed consent.
* Healthy females and males aged 18 - 55 years .
* No clinically significant health problems
* Body mass index 18.5 - 30.0 kg/m2 and weight >50 kg at screening.
* Females of childbearing potential who agree to comply with the applicable contraceptive requirements of the protocol or females who are permanently sterilized.
* Males who agree to comply with the applicable contraceptive requirements of the protocol
* Subjects must be willing to minimize blood and body fluid exposure of others for 7 days after vaccination
* Be willing to refrain from blood donation during the course of the study.
* The subject is co-operative and available for the entire study.

Exclusion Criteria:

* Prior receipt of an Ebolavirus or Marburgvirus vaccine or VSV-vectored vaccine.
* Receipt of any vaccine in the 2 weeks prior to the trial vaccination (4 weeks for live vaccines) or planned receipt of any vaccine in the 3 weeks following the trial vaccination.
* Known allergy to the components of the BPSC1001 vaccine product or history of life-threatening reactions to vaccine containing the same substances.
* Participation in a clinical trial or use of an investigational product within 30 days or five times the half-life of the investigational drug -prior to receiving the first dose within this study
* Evidence in the subject's medical history or in the medical examination that might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the investigational product under investigation.
* Any positive result for HIV1/2, HCV antibody or HBs antigen testing.
* Pregnant or lactating females, or females who intend to become pregnant during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or diabetes
* Subjects with inflammatory, infectious and neuroinflammatory underlying disease which could cause an expected impairment of the blood brain barrier such as meningitis, multiple sclerosis, epilepsy, or Alzheimer's.
* Any household contact who is immunodeficient, HIV positive or pregnant
* Working with livestock
* Any chronic or active neurologic disorder, including migraines, seizures, and epilepsy, exclud-ing a single febrile seizure as a child
* Known history of Guillain-Barré Syndrome
* Active malignancy or history of metastatic or hematologic malignancy
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years
* Moderate or severe illness and/or fever >38°C within 1 week prior to vaccination
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* History of blood donation within 60 days of enrollment or plans to donate within the study period
* Receipt of chronic immune suppressants or other immune-modifying drugs within 6 months of study inclusion
* Subjects with skin lesions close to the injection site or active oral lesions will be excluded.
* Thrombocytopenia, contraindicating intramuscular vaccination based on investigator's judgment
* Subjects with a significant infection or known inflammation.
* History of relevant cardiovascular disorders or evidence of hyper- or hypotension
* Subjects who are known or suspected not to comply with the study directives.
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The number of adverse events associated with the rVSVΔ-ZEBOV-GP (BPSC1001) vaccine will be collected and measured | Vaccination (day 0) to day 180

SECONDARY OUTCOMES:
ZEBOV-GP-specific antibody responses | Vaccination (day 0) to day 180
  Humoral immunity: Magnitude of ZEBOV-GP-specific antibody responses as assayed by ELISA in a centralized laboratory.
To evaluate vaccine viremia and excretion | Vaccination (day 0) to day 28
  Vaccine viremia and viral shedding: concentration of rVSV in peripheral blood, urine and saliva as detected by qRT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M. Addo, MD, Study Director — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- CTC North GmbH & Co. KG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poetsch JH, Dahlke C, Zinser ME, Kasonta R, Lunemann S, Rechtien A, Ly ML, Stubbe HC, Krahling V, Biedenkopf N, Eickmann M, Fehling SK, Olearo F, Strecker T, Sharma P, Lang KS, Lohse AW, Schmiedel S, Becker S; VSV-Ebola Consortium (VEBCON); Addo MM. Detectable Vesicular Stomatitis Virus (VSV)-Specific Humoral and Cellular Immune Responses Following VSV-Ebola Virus Vaccination in Humans. J Infect Dis. 2019 Jan 29;219(4):556-561. doi: 10.1093/infdis/jiy565. PMID 30452666
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166
- [Derived] Dahlke C, Kasonta R, Lunemann S, Krahling V, Zinser ME, Biedenkopf N, Fehling SK, Ly ML, Rechtien A, Stubbe HC, Olearo F, Borregaard S, Jambrecina A, Stahl F, Strecker T, Eickmann M, Lutgehetmann M, Spohn M, Schmiedel S, Lohse AW, Becker S, Addo MM; VEBCON Consortium. Dose-dependent T-cell Dynamics and Cytokine Cascade Following rVSV-ZEBOV Immunization. EBioMedicine. 2017 May;19:107-118. doi: 10.1016/j.ebiom.2017.03.045. Epub 2017 Apr 5. PMID 28434944
- [Derived] Medaglini D, Harandi AM, Ottenhoff TH, Siegrist CA; VSV-Ebovac Consortium. Ebola vaccine R&D: Filling the knowledge gaps. Sci Transl Med. 2015 Dec 9;7(317):317ps24. doi: 10.1126/scitranslmed.aad3106. PMID 26659569
- [Derived] Agnandji ST, Huttner A, Zinser ME, Njuguna P, Dahlke C, Fernandes JF, Yerly S, Dayer JA, Kraehling V, Kasonta R, Adegnika AA, Altfeld M, Auderset F, Bache EB, Biedenkopf N, Borregaard S, Brosnahan JS, Burrow R, Combescure C, Desmeules J, Eickmann M, Fehling SK, Finckh A, Goncalves AR, Grobusch MP, Hooper J, Jambrecina A, Kabwende AL, Kaya G, Kimani D, Lell B, Lemaitre B, Lohse AW, Massinga-Loembe M, Matthey A, Mordmuller B, Nolting A, Ogwang C, Ramharter M, Schmidt-Chanasit J, Schmiedel S, Silvera P, Stahl FR, Staines HM, Strecker T, Stubbe HC, Tsofa B, Zaki S, Fast P, Moorthy V, Kaiser L, Krishna S, Becker S, Kieny MP, Bejon P, Kremsner PG, Addo MM, Siegrist CA. Phase 1 Trials of rVSV Ebola Vaccine in Africa and Europe. N Engl J Med. 2016 Apr 28;374(17):1647-60. doi: 10.1056/NEJMoa1502924. Epub 2015 Apr 1. PMID 25830326